CLINICAL TRIAL: NCT03693729
Title: Effects of Brain-stimulation on Memory and Memory Awareness
Brief Title: Effects of Brain-stimulation on Metamemory Monitoring and Control
Acronym: FOKhint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brooklyn College of the City University of New York (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Chua, Associate Professor, Brooklyn College of the City University of New York
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BrooklynC; SC3GM121192 (NIH)
Record Dates: First submitted 2018-09-21; First posted 2018-10-03 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: memory; metacognition; metamemory; transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active DLPFC during task (Experimental): HD-tDCS will be applied over the DLPFC at 2mA in a single session for up to 30 min during the memory and metamemory task
  Interventions: Device: HD-tDCS
- Active DLPFC after task (Active Comparator): HD-tDCS will be applied over the DLPFC at 2mA in a single session for up to 30 min after the memory and metamemory task and during a filler task.
  Interventions: Device: HD-tDCS
- Sham DLPFC during task (Sham Comparator): Sham HD-tDCS will be applied over the DLPFC at 2mA in a single session for up to 30 min during the memory and metamemory task
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — Participants will complete a metamemory and memory task
  Other Names: Behavioral

SUMMARY:
When people learn and remember information, it is often accompanied by a feeling of subjective confidence about whether or not information has been learned and accurately remembered. These subjective feelings of confidence are often related to actual memory performance, but are sometimes incorrect. The investigators have previously shown that applying high definition transcranial direct current stimulation (HD-tDCS) over the dorsolateral prefrontal cortex leads to more accurate feelings of subjective confidence, at least when subjects are asked for their confidence about future memory performance. Accurate confidence judgments are useful in that they may later subsequent behavior, and inaccurate ones may be costly. For example, a student who erroneously believes that studied material was learned may stop studying and not do well on a test. Individuals who have a feeling-of-knowing about the answer to a general knowledge question will continue to search their memory, whereas individuals who do not have a feeling-of-knowing will stop searching their memory. Individuals who are confident they know the answer to a question are more likely to answer it. In this study, the experimenters are testing the effects of brain stimulation on subjective awareness of memory (termed metamemory monitoring) and how people use those subjective judgments (termed metamemory control). The approach taken is to have participants visit the laboratory on 3 visits and receive brain stimulation while completing memory and metamemory tasks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, right-handed adults ages 18-35. English spoken since age 5. Normal or corrected-to-normal vision.

Exclusion Criteria:

* Participants will be excluded if they have chronic skin disease or a medical skin condition, or an unhealed open wound on the scalp, face, neck, or forehead near the electrode location.
* Participants will be excluded if they self-report significant medical, neurological, or psychiatric illness and/or a history of substance abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Memory Control Advantage Index | Through study completion, an average of 3 weeks
  This indexes the memory advantage for choosing which general knowledge question one receives a hint about the answer to versus having the experimenter choose which general knowledge question one receives a hint about the answer. The investigators will subtract the proportion of correctly recognized general knowledge answers for experimenter-chosen questions from the proportion correctly recognized for participant-chosen questions

SECONDARY OUTCOMES:
semantic recognition as assessed by a general knowledge task | Through study completion, an average of 3 weeks
  Differences in recognition are compared between each condition (each active HD-tDCS and sham).
semantic recall as assessed by a general knowledge task | Through study completion, an average of 3 weeks
  Differences in recall are compared between each condition (each active HD-tDCS and sham).
Feeling-of-knowing ratings and their accuracy | Through study completion, an average of 3 weeks
  Feeling of knowing ratings are given on a scale. To assess the accuracy of these ratings, the subjective ratings are compared to objective accuracy, using signal detection based measures. Differences in feeling-of-knowing ratings and their accuracy are compared between each condition (each active HD-tDCS and sham).

CONTACTS AND LOCATIONS:
Locations (1):
- Brooklyn College, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided